CLINICAL TRIAL: NCT07130409
Title: Multimodal Imaging Assessment After Revascularization in Patients With Acute Myocardial Infarction
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Other Study IDs: QYFYECR2025-74
Record Dates: First submitted 2025-07-30; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Magnetic Resonance Imaging; Acute Myocardial Infarction (AMI); PET / MR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- clinically diagnosed with first-episode AMI and undergoing interventional therapy

SUMMARY:
This prospective cohort study will enroll 20 patients clinically diagnosed with first-time acute myocardial infarction (AMI) who underwent interventional procedures (including percutaneous coronary intervention [PCI] and balloon angioplasty) at the Affiliated Hospital of Qingdao University. Patient data, including routine blood and urine tests, blood biochemistry, electrocardiograms (ECG), imaging studies, and interventional procedure records, will be collected to assess eligibility for enrollment. The study procedures include patient screening and enrollment, obtaining informed consent, baseline assessment (including medical history, laboratory tests, ECG, etc.), an ¹⁸F-Pentixafor PET/MR examination, and follow-up. Images will be blindly assessed by at least two specialized physicians from the Radiology and Nuclear Medicine departments. The study aims to investigate the utility of ¹⁸F-Pentixafor PET/MR in evaluating coronary microcirculatory function, cardiac function, myocardial viability, myocardial inflammatory response, and the efficacy of interventional therapy in AMI patients post-procedure. Additionally, it will perform risk stratification and prognostic analysis for the enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of first-episode acute myocardial infarction (AMI) who underwent emergency percutaneous coronary intervention (PCI) were included. All patients had complete baseline clinical data, with baseline cardiac magnetic resonance (CMR) examinations performed within 7 days post-PCI and follow-up CMR completed at 6 months post-procedure.

Exclusion Criteria:

* Patients with severe cardiac decompensation (Killip class 4) or clinically unstable conditions.

Patients with coexisting valvular heart disease, congenital heart disease, pulmonary hypertension, cardiomyopathy, or persistent atrial fibrillation that may confound cardiac structural/functional assessments.

Prior history of myocardial infarction, coronary revascularization (PCI/CABG).

Concurrent severe systemic diseases including hematologic disorders, malignancies, rheumatic/autoimmune diseases, or severe hepatic/renal failure.

Contraindications to CMR (claustrophobia, pacemaker implantation, etc.).

Pregnant, breastfeeding, or women of childbearing potential without effective contraception.

Sexually active individuals of reproductive age unwilling to use reliable contraception.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clinically diagnosed with first-episode AMI and undergoing interventional therapy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The myocardial uptake of 18F-Pentixafor was quantified using SUVmax and SUVmean values derived from PET imaging. | At baseline (within 1 week of enrollment)
Left ventricular ejection fraction (LVEF) assessed by cardiac MRI to evaluate left ventricular function | At baseline (within 1 week of enrollment)
Infarct Characterization | At baseline (within 1 week of enrollment)
  Late gadolinium enhancement (LGE) images were used to calculate infarct size (IS).

SECONDARY OUTCOMES:
Myocardial T1 Values and Extracellular Volume (ECV) | At baseline (within 1 week of enrollment)
  Myocardial T1 values within the LGE territory were measured to yield native T1 and post-contrast T1 values. ECV was calculated using the native and post-contrast myocardial T1 values, blood pool T1 values, and the hematocrit (HCT).
Myocardial T2 values | At baseline (within 1 week of enrollment)
  Myocardial T2 values were quantified using T2 mapping images to assess myocardial edema.
Myocardial Strain Analysis | At baseline (within 1 week of enrollment)
  Feature-tracking analysis (CMR-FT module, CVI42) was performed offline on cine sequences. LV endocardial and epicardial contours were automatically tracked at end-diastole and end-systole, followed by manual adjustments as necessary. Global and segmental myocardial strain values were derived.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No